CLINICAL TRIAL: NCT01944579
Title: Blackberry Flavonoid Absorption and Effects on Intestinal Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janet Novotny (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: HS40
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control-Blackberry (Experimental): Participants will receive a controlled diet with the control food (jello) first and then cross over to the controlled diet with blackberries.
  Interventions: Other: Blackberries; Other: Control
- Blackberry-Control (Experimental): Participants will receive a controlled diet with blackberries first and then cross over to the controlled diet with the control food (jello).
  Interventions: Other: Blackberries; Other: Control

INTERVENTIONS:
Other: Blackberries — Participants will receive blackberries as part of a controlled diet.
Other: Control — Participants will receive a control food (jello) as part of a controlled diet.

SUMMARY:
Intestinal bacteria can metabolize unabsorbed polyphenols (plant compounds) to produce smaller molecules which may impact health. In addition, evidence suggests that this process may be affected by body fatness. This study aims to investigate absorption of blackberry polyphenols, their impact on intestinal bacteria, polyphenol metabolites formed by intestinal bacteria, and how these processes differ for obese and lean individuals. It is hypothesized that polyphenol absorption and metabolism will differ between obese and lean individuals and that differences in intestinal microbiota may play a role.

ELIGIBILITY:
Inclusion Criteria:

* 25-75 years old

Exclusion Criteria:

* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol (dicumarol), or Miradon (anisindione)
* Presence of any gastrointestinal disease, metabolic disease, or malabsorption syndromes that may interfere with the study goals
* Have been pregnant during the previous 12 months, are currently pregnant or lactating, or plan to become pregnant during the study
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* Fasting triglycerides greater than 300 mg/dL
* Fasting glucose greater than 126 mg/dL
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanolamine, ephedrine, caffeine) during and for at least 6 months prior to the start of the study or a history of a surgical intervention for obesity
* Active cardiovascular disease (such as a heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within the last three months, stroke, or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in the past six months).
* Use of any tobacco products in past 3 months
* Unwillingness to abstain from herbal supplements for two weeks prior to the study and during the study
* Known (self-reported) allergy or adverse reaction to blackberries or other study foods
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past twelve months and/or current acute treatment or rehabilitation program for these problems (Long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in fecal microbiota | 0 weeks, 4 weeks
  Feces will be analyzed for bacterial typing at 0 and 4 weeks of each diet period.

SECONDARY OUTCOMES:
Change in blackberry nutrients & metabolites | 0, 30, 60, 90, 120, 150, 180, 240, 300, 360, and 420 minutes

OTHER OUTCOMES:
Change in gene expression | 0 weeks, 4 weeks
  Gene expression in whole blood will be evaluated at the beginning and end of each diet period, through global gene expression using the Affymetrix platform. Changes in specific genes observed with global gene expression technology will be confirmed through RT-PCR.
Change in metabolomics | 0 weeks, 4 weeks
  Blood, urine, and feces will be analyzed by a technique called metabolomics, which is a broad sampling of metabolites.
Change in biomarkers of cancer | 0 weeks, 4 weeks
  Biomarkers of cancer risk such as oxidative stress and inflammatory markers will be analyzed at the beginning and end of each diet period.
Change in lipopolysaccharide | 0 weeks, 4 weeks
  Lipopolysaccharide will be measured in the blood as a measure of gut leakiness.

CONTACTS AND LOCATIONS:
Overall Officials: Janet A Novotny, Ph.D., Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States